CLINICAL TRIAL: NCT01322061
Title: The Role of a Single Oral Dose (2g) of Vitamin C in Reducing Intensity of Pain and Opioids Consumption in Patients Undergoing Laparoscopic Cholecystectomy. A Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Vitamin C Efficacy in Reducing Post Operative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ghassan Kanazi, Associate Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES.GK.06; AUBMC (Other: AUBMC)
Record Dates: First submitted 2011-03-09; First posted 2011-03-24 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Gallbladder Inflammation
Keywords: Gallbladder removal; acute cholecystitis; Laparoscopic cholecestectomy
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin C (Active Comparator)
  Interventions: Drug: Ascorbic Acid
- mirinda (Placebo Comparator)
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Effervescent,1000mg/tablet, 2000 mg dissolved in 50ml water, the drug will be given once, one hour prior to surgery
  Other Names: Redoxon, Vitamin C 1000mg, Bayer LSR912 MFD

SUMMARY:
Opioids are the corner stone in the treatment of post operative pain. Because of the several side effects of opiods, non-steroidal anti-inflammatory drugs are usually added postoperatively to decrease the total requirements of opioids. However, non steroidal anti-inflammatory drugs have side effects of their own. Vitamin C, with virtually no side effects when used on short-term basis, has been shown to have promising analgesic effects in chronic pain and acute pain relief following orthopedic surgeries.

The investigators propose to assess the role of a prophylactic single dose (2g) of vitamin C in reducing the intensity of pain and the consumption of opioids in patients undergoing laparoscopic cholecystectomy at AUB-MC.

All eligible patients undergoing laparoscopic cholecystectomy at AUB-MC will be included in the study. Patients will be randomized into two groups to receive either single dose oral vitamin C (2g) (Study Group) or identically looking placebo capsules (Control Group). Both the patients and the investigation team will be blinded to the type of intervention. Intraoperative anesthesia management will be similar for both groups. Postoperative pain control will be achieved with patient controlled analgesia via a patient controlled morphine pump in both groups. At several time intervals and up to 24 hours postoperatively, the pain scores, morphine consumptions, nausea/vomiting scores, sedation scales, itching scales, and patient satisfaction scales will be obtained for all patients. Also, the peak vitamin C concentration will be determined for each patient.

Patients demographics will be obtained and compared between both groups. The differences in pain scores, morphine consumptions, nausea/vomiting scores, and sedation, itching, and patient satisfaction scales will be compared between the two groups with the Student-t test, the analysis of variance, the Fisher exact test, and the Kruskal-Wallis test. The peak vitamin C plasma concentration will be correlated with the pain scores in each group using regression analysis.

This study will provide relevant information on whether a single dose (2g) of vitamin C can reduce morphine requirements and non steroidal anti-inflammatory drugs need and thus eliminating their side effects in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender
* Between 18-75 years old
* ASA class I, II, or III
* Scheduled to undergo laparoscopic cholecystectomy

Exclusion Criteria:

* Intake of anti-inflammatory drug in the past 24 hr
* Allergy to morphine
* History of chemical dependence
* Chronic pain state
* Inability to use PCA pumps
* History of obstructive sleep apnea
* History of severe asthma
* History of COPD
* History of gastroesophageal reflux disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | total morphine consumption in 24 hours
  During their stay in the PACU (Post Anesthesia Care Unit), patients in both groups will be started on a morphine IV PCA pump that is programmed to deliver on patient's demand 1mg every 6 minutes with a total limit of 30mg every 4 hours for post operative relief.Patients will be followed up after discharge from PACU and morphine consumption will be recorded

SECONDARY OUTCOMES:
sedation score on the Ramsey scale | Sedation score will be measured in PACU and up 24 hours upon discharge from PACU
incidence of nausea and vomiting | Nausea and vomiting incidence will be monitored in PACU and up 24 hours upon discharge from PACU
  Nausea/Vomiting will be monitored using Verbal Rating Score (VRS). The number of vomiting episodes will be recorded. Episodes of vomiting occurring less than 5 min-apart will be considered as one episode.
Incidence of itching | Itching incidence will be measured in PACU and up 24 hours upon discharge from PACU
patient satisfaction scale | patient satisfaction scale will be measured in PACU and up 24 hours upon discharge from PACU
  Patient satisfaction scale measures the overall patient's satisfaction regarding the post-operative experience in terms of pain managment. The scale is divided into four main categories: Excellent, Good, Fair,Poor.
Pain score on the Visual Analog Scale | Pain will be measured in PACU and up to 24 hours upon discharge from PACU
  During their stay in the PACU, the incisional, visceral and shoulder pain intensity for each patient will be measured using Visual Analog Scale (VAS)and/or Verbal Rating Score.

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Kanazi, MD, Principal Investigator — AUBMC
Locations (1):
- AUBMC, Beirut, Beyrouth, Lebanon

REFERENCES:
- [Derived] Kanazi GE, El-Khatib MF, Yazbeck-Karam VG, Hanna JE, Masri B, Aouad MT. Effect of vitamin C on morphine use after laparoscopic cholecystectomy: a randomized controlled trial. Can J Anaesth. 2012 Jun;59(6):538-43. doi: 10.1007/s12630-012-9692-x. Epub 2012 Mar 9. PMID 22402954